CLINICAL TRIAL: NCT02832401
Title: The Impact of Caffeine on Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other); Mount Saint Vincent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1021504
Record Dates: First submitted 2016-06-30; First posted 2016-07-14 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia; Caffeine
Keywords: event-related potentials; EEG; caffeine; psychosis; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Active Comparator): 200 mg of caffeine powder administered in capsules
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Cellulose powder administered in capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine
  Arms: Caffeine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Caffeine is the most used psychoactive drug in Canada, with regular consumption by 88% of the adult population, While rates of caffeine consumption are considered to be high in the general population, there is some evidence that they may be even higher within schizophrenia patients; in a 2006 U.S. study, daily consumption rates of caffeine were nearly double those observed in a healthy control population (471.6 mg/day vs. 254.2 mg/day). Furthermore, 13% of the schizophrenia population studied ingested more than 1000 mg/day of caffeine, well above the 400 mg daily maximum recommended by Health Canada. High doses of caffeine are particularly concerning for individuals with schizophrenia; caffeine alters dopaminergic activity at post-synaptic neurons through its actions at adenosine A2A receptors, which may exacerbate positive symptoms, such as delusions and hallucination. This significant rate of consumption is likely due in part to caffeine's actions on the human brain, resulting in increased arousal, elevated mood and beneficial effects on a wide-range of cognitive processes including verbal working memory, sustained attention, and executive function. These areas of caffeine-induced cognitive improvement notably overlap with the cognitive domains that are reported to be diminished in schizophrenia. Despite this overlap and the rates of caffeine consumption observed within schizophrenia, research reports examining the effects of caffeine on cognition and brain activity are all but non-existent in this population. The primary objective of this proposal is to compare the effects of caffeine and placebo on brain function during cognitive tasks in participants with schizophrenia. While the investigators have specific hypotheses for each task, overall the investigators hypothesize that caffeine will improve cognitive function (as evidenced by larger ERP amplitudes and/or reduced ERP latencies) compared to placebo in schizophrenia patients, with similar effects (albeit reduced in magnitude) observed in non-patient healthy controls.

DETAILED DESCRIPTION:
1.1 Background. Caffeine is the most used psychoactive drug in Canada, with regular consumption by 88% of the adult population and is unique because it is a "cradle-to-grave drug". In Canada, coffee is the most commonly consumed source of caffeine, while tea, chocolate and energy drinks are also significantly used. This significant rate of consumption is likely due in part to caffeine's actions on the human brain, resulting in increased arousal, elevated mood and cognitive enhancements. The effects of caffeine, at least at levels typically seen in human consumption, are primarily related to its actions at adenosine receptors. Caffeine's antagonistic effects on adenosine can be seen after even a single cup of coffee, with increased consumption resulting in increased blockade. Adenosine receptors are distributed in all brain cells, contributing to the caffeine's ability to affect a wide range of brain regions.

While levels of caffeine consumption are considered to be high in the general population, there is some evidence that they may be even higher within schizophrenia (SZ) patients. In a recent U.S. study of 146 community-dwelling individuals with SZ, daily consumption rates of caffeine were nearly double those observed in a healthy control population (471.6 mg/day vs. 254.2 mg/day; p < .001). Furthermore, 13% of the SZ population studied ingested more than 1000 mg/day of caffeine, with the highest observed intake at 2647.2 mg/day. To place this in context, Health Canada recommends adults consume no more than 400 mg of caffeine per day, and doses above 250 mg have the potential to induce symptoms of anxiety, agitation, irritability and insomnia . High doses of caffeine are particularly concerning for individuals with SZ as caffeine alters dopaminergic activity at post-synaptic neurons through its actions at adenosine A2A receptors; this enhances dopamine function, resulting in increased locomotor activity and appears to exacerbate positive symptoms, such as delusions and hallucinations . Another effect of caffeine with particular relevance to SZ involves its interaction with atypical antipsychotic drugs, such as clozapine. Both clozapine and caffeine are metabolized in the liver by the cytochrome P450 system and, in particular, the CYP1A2 isoenzyme. Competition between clozapine and caffeine has been reported to elevate antipsychotic blood levels, increasing the risk of clinically significant side effects at high dosage levels of caffeine. As such, given the high consumption levels and potential negative side effects of caffeine in SZ, it is important to understand the cortical mechanisms that underlie caffeine use.

As caffeine is mainly used because of perceived stimulant properties, including enhanced mental alertness and increased energy, research has been conducted to examine the effects of caffeine on cognitive performance in humans. These studies have identified beneficial effects of caffeine on a wide-range of cognitive processes including verbal working memory, sustained attention, and executive function. It must be noted, however, that while many studies report pro-cognitive effects of caffeine, others report no significant improvements or deficits in performance. This may be at least partially explained by evidence suggesting an 'inverted U-shaped' dose-response curve for caffeine, wherein lower doses have positive effects on performance, while high doses (i.e., above 500 mg) cause a decrease in performance.

Within the fields of attention and information processing, the electroencephalographically (EEG)-derived event-related potentials (ERPs) provide an exquisitely sensitive method of indexing cognition that can both complement and clarify behavioural observations. The ERP waveform is elicited in response to a specific stimulus, such as tones or light flashes, or cognitive events, such as recognition, decision making or response to specific stimuli events. Specifically, ERPs represent an average of the neural activity that follows the onset of a stimulus. In studies examining the effects of caffeine on the brain, EEG/ERPs appear to be preferable to neuroimaging techniques such as fMRI and PET as the vasoconstrictive nature of caffeine may confound these latter techniques, which model cortical blood flow. EEG/ERPs avoid these potential confounds and, furthermore, provide a temporal resolution far superior to some of the more sophisticated imaging techniques (i.e. PET, fMRI), making this methodology far more suitable for capturing instantaneous changes in information processing. While the literature of caffeine's effects on ERP-indexed cognitive processes is limited, there is evidence of caffeine enhancing ERPs. In one such study, not only was there quicker behavioural responding during a visual search task with caffeine (vs. placebo), but also quicker ERP measures of target detection, although caffeine did not alter ERP amplitudes.

While a hallmark characteristic of SZ is neurocognitive impairment, these deficits notably overlap with the cognitive domains that are improved by caffeine. Among the core deficts observed within SZ is a dysfunction of attentional systems, which can be observed in patients who are both acutely psychotic and in remission. Deficits of attention in SZ include both alteration of sustained attention, particularly as measured by continuous performance tasks and visual selective attention (Luck & Gold, 2008), as measured by visual search tasks. It has further been suggested that within SZ these deficits of attention contribute to dysfunction of the central executive and working memory, the limited capacity system for storing and manipulating information for short time periods (up to ~30 s), in order to carry out complex cognitive operations such as planning, reasoning, and problem solving. Impairment in working memory processes, such as those indexed by the n-back task, are a robust feature of SZ, are stable over time, and independent of psychotic symptoms.

While there is a literature, albeit small, examining the effects of caffeine on cognition and brain activity in healthy individuals, such research reports are all but non-existent in SZ (based on extensive searches with both PsycINFO and PubMed). This gap in the literature is particularly notable given the rates of caffeine consumption observed within SZ. The sole studies to address how caffeine might impact cognitive processes in SZ have done so within animal models employing MK-801 (a potent NMDA receptor antagonist) infused mice. Within this behavioural model of SZ, chronic treatment with caffeine improved measures of long term memory, while reducing MK-801-induced perseverative errors in one study, while another study found no effects of chronic caffeine on cognition in mice given a significantly higher dose of MK-801.

1.2 Objective. This project proposes to examine how caffeine alters ERP-indexed aspects of cognition in SZ patients. Neural (ERPs) and behavioural (hits, reaction time) correlates of cognitive performance will be probed within a randomized, double-blind, placebo-controlled design with a battery of well-established cognitive paradigms that have both demonstrated deficits in SZ and are associated with caffeine-induced enhancement: a visual selective attention paradigm (visual search task), a working memory paradigm (N-back), and a sustained attention paradigm (AX-CPT). The primary outcome measures will be ERP amplitudes and latencies. Secondary indices will include behavioural measures of performance, including accuracy (% correct), reaction times and measures of signal detection (i.e. d'). While the investigators expect caffeine to improve behavioural and neural indices in both groups, the investigators expect this effect to be stronger in SZ patients due to expected lower baselines.

2. Materials and Methods. 2.1 Study Design and Procedure. This study will employ a randomized, placebo-controlled, double-blind, repeated measures design consisting of two experimental sessions separated by at least 24 hrs, with participants receiving caffeine one day and placebo on the other day. The order of caffeine administration will be counterbalanced, such that half of the participants are randomly administered caffeine in the first and placebo in the second session, while the remaining half are administered caffeine and placebo in the reverse order. Prior to the experimental sessions, participants will complete informed consent, having been given an opportunity to read the study description and have any questions answered, complete demographic questionnaires, and experimental sessions will be scheduled. Participants will attend the BIOTIC Neuroimaging Research Lab at the QEII Health Sciences Centre (Halifax, NS), for a morning (i.e. testing beginning between 9-11 am) testing session. Participants will be required to abstain from illicit drugs, over-the-counter medications, alcohol and cigarettes beginning at midnight of the previous day. SZ patients will not be asked to halt or pause any current medication regimen. Additionally, participants will be asked to abstain from caffeine (including coffee, tea and cola) for at least 6 hours prior to the test session to ensure adequate clearance of circulating caffeine (half-life = 2.5-4.5 hrs). Upon arrival at the laboratory, following self-report of adherence to pre-testing abstinence, drug treatment will be administered, EEG electrodes will be applied and, 30 minutes after drug administration, volunteers will be assessed with the test battery, presented in a randomized order to avoid order effects. All testing procedures will be carried out in accordance with the Declaration of Helsinki and following the approval of the relevant research ethics boards.

2.2 Caffeine. As in previous studies investigating the effects of caffeine on electrophysiological measures, in each session participants will be asked to swallow (with water) one of two identical pill capsules containing either caffeine (200 mg) or placebo. This method and dosage were selected as oral administration of caffeine results in efficient absorption, while the intermediate size dose, which is typical of most studies of caffeine on cognition, has been shown to exert widespread, strong cerebral effects. Furthermore, administration of caffeine in pill form allows for greater control over dosage and facilitates double-blind procedures, while controlling for potentially confounding sensory effects (e.g. smell, taste of coffee).

2.3 Test Battery. 2.3.1 Visual Search Task. The visual search task will follow methodology described by Lorenzo-Lopez and colleagues and previously used in psychopharmacology research. In short, participants will be instructed to perform a visual search, which consists of detecting a target stimulus (vertical bar) among an array of distractors (horizontal bars) by indicating whether the target was present or absent in each search array by pressing a green button on a response pad with one hand and a red button with the other hand, respectively. Behavioral measures will include the number of correct responses, and the reaction times (RTs) of correct responses. Neural (ERP) measures of interest include the N2pc, an index of visual spatial shifts of attention to the location of the target or distractor, and the P3b, an index of target detection. The amplitudes of these ERPs indicate the amount of resources allocated to the associated cognitive process, while latency represents processing speed. Hypotheses: Caffeine will significantly speed up behavioural indices of target detection (i.e. reduced RTs) and associated neural waveforms (i.e. reduced latency of N2pc & P3b) in both groups, with an increase in amplitude only observed in SZ patients.

2.3.2 Visual Sustained Attention (AX-CPT). Sustained attention will be assessed within the A-X version of the continuous performance task (AX-CPT). Participants will be presented with a series of letters and will be instructed to respond to the letter "X" only when it was immediately preceded by "A." In order to test sustained attention, 400 letters will be presented over a span of 11 minutes consisting of 80 cues ("A"), 40 targets ("A" followed by "X"), 40 NoGos ("A" followed by any other letter), and 240 distractors (other letters or "X" not preceded by "A"). Behavioural endpoints include the number and RTs of correct responses, and false alarms (i.e., nontarget responses). Neural (ERP) measures of interest include the P3b to correct targets. Hypotheses: Consistent with previous reports in sustained attention, caffeine will not impact behavioural performance, but will increase P300 amplitudes, with this effect (vs. placebo) being seen in both participant groups.

2.3.3 Visual Working Memory. This paradigm, which has previously been used in psychopharmacology research, will employ four randomized conditions of the verbal N-Back task; each condition will have identical stimuli and response demands, but consist of increasing levels of working-memory load. A series of letters will be presented and participants will be required to respond as quickly as possible only when the letter on the screen matches the letter n stimuli back (i.e., for the 0-back condition, the target is any letter that matches a pre-specified letter (x), while in the 1-back, 2-back and 3-back conditions, a target is any letter that is identical to the letter presented one, two or three trials back, respectively). As the N-back task requires information storage, updating, and manipulation, it has become the dominant tool used in assessing WM control functions. Behavioural endpoint measures will include accuracy (% correct target detections) and reaction time (ms) to targets. Additionally, for each condition and each drug treatment I will calculate signal detection sensitivity (d') and response bias (C). Electrophysiological endpoint measures include amplitudes and latencies of the P3b to targets. Hypotheses: Similar to the other paradigms, and consistent with behavioural studies of caffeine's effects on n-back indexed working memory, the investigators expect caffeine will reduce RTs and will reduce P300 latency in both groups.

2.4 EEG Recording and ERP Computation. ERPs will be extracted from EEG activity recorded from an electrode cap with Ag+/Ag+-Cl- active electrodes at sixty-four scalp sites according to the 10-10 system of electrode placement, including: three midline sites (frontal [Fz], central [Cz], parietal [Pz]); three left hemisphere (frontal [F3], central [C3], parietal [P3]) and three right hemisphere (frontal [F4], central [C4], parietal [P4]) scalp sites; and bilateral mastoid activity. Electrodes will be also placed on the mid-forehead and nose to serve as ground and reference, respectively. Bipolar recordings of horizontal (HEOG) and vertical (VEOG) electro-oculogram activity will be taken from supra-/sub-orbital and external canthi sites, respectively. All electrode impedances will be kept below 5kohms. Electrical activity will be recorded with an amplifier bandpass of 0.1 and 30 Hz, digitized at 500 Hz, and stored on hard-disk for later off-line analysis. Stimuli (and resulting triggers for ERP analysis) will be generated by Presentation software (Neurobehavioural Systems, Berkeley CA) 2.5 Questionnaires. In order to assess clinical variables in SZ patients, as well as caffeine consumption, 2 questionnaires will be administered: 1) Psychotic Symptom Rating Scale (PSYRATS). The PSYRATS is designed to quantify auditory hallucinations and delusions, both of which have been associated with consumption of caffeine; 2) Caffeine Consumption Questionnaire (CCQ). Collects detailed information on caffeine consumption, including sources of caffeine (e.g., coffee, cola, etc…) and time period of caffeine consumption. As both of these questionnaires probe trait (vs. state) measures, they will only be administered once.

2.6 Data Analysis. Data will be subjected to separate ANOVA/ANCOVA procedures (SPSS, IBM Corp., Armonk NY). For each paradigm, endpoint measures will be analyzed by mixed ANOVAs, with between-group (2 levels: patients, controls) and within-group/repeated measures factors including drug (caffeine, placebo). Analysis of EEG/ERP endpoints will also include scalp site as a within-group factor. Daily caffeine consumption (as measured by the CCQ) will be used as a covariate. Follow-up of significant (Greenhouse-Geisser corrected) main or interaction effects (p < .05) will be carried out with Bonferroni-adjusted planned comparisons using separate (vs. pooled) error estimates. In order to examine the correlation between behavioural/electrophysiological endpoints and measures of caffeine consumption, two-tailed Spearman's rho correlations will be conducted between consumption measures and ERP amplitudes/latencies under placebo and drug conditions, as well as between consumption measures and measures of drug-associated change in ERP endpoints overall and within both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants: Patients will have a primary diagnosis of schizophrenia and will be judged as clinically stable, as indicated by the patient's primary physician and including no changes in symptoms or antipsychotic medications for the last 2 months, and each participant's primary medication (if any) will be limited to one of the atypical anti-psychotics, excluding clozapine due to the noted interactions. Participants will be required to understand spoken and written English and will be right-handed (assessed by the Edinburgh Handedness Inventory [EHI]) to facilitate source localization techniques. Participants will be required to have normal (or corrected) vision.
* Healthy controls: Self-report of negative psychiatric, medical, neurological and alcohol/drug abuse histories, and current non-use of medications (with the exception of oral contraceptives). Participants will be required to understand spoken and written English and will be right-handed (assessed by the Edinburgh Handedness Inventory [EHI]) to facilitate source localization techniques. Participants will be required to have normal (or corrected) vision.

Exclusion Criteria:

* Patients: Patient participants will be excluded if they meet any of the following criteria: co-morbid DSM-IV TR Axis I disorder; current treatment with clozapine; total PANSS score >65, reflecting an acute psychotic episode; current history of drug abuse or dependence; history of head injury resulting in loss of consciousness; diagnosis of epilepsy or any other neurologic disorder; electro-convulsive therapy (ECT) treatment within the previous year; significant cardiac illness; or extrapyramidal symptoms (EPS) resulting in movement disorders which could affect ERP recordings. Additionally, as is common in caffeine research, participants will be excluded if they work night shifts or do not report normal (i.e. nocturnal) sleep patterns during screening
* Healthy Controls: As is common in caffeine research, participants will be excluded if they work night shifts or do not report normal (i.e. nocturnal) sleep patterns during screening.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Event-related potentials (ERPs) | 30 minutes post-intervention during both test sessions
  Average neuroelectric brain response measured in microvolts. Event-related potentials include N2pc (visual search) and P300 (visual search, AX-CPT and N-Back)

SECONDARY OUTCOMES:
Response accuracy | 30 minutes post-intervention during both test sessions
  % of correct responses during performance of visual search, AX-CPT and N-Back
Reaction Time | 30 minutes post-intervention during both test sessions
  Average time from target appearance to correct behavioural response (measured in milliseconds) during performance of visual search, AX-CPT and N-Back
False alarms | 30 minutes post-intervention during both test sessions
  Number of responses to non-target stimuli during performance of visual search, AX-CPT and N-Back
d' | 30 minutes post-intervention during both test sessions
  A measure of signal detection sensitivity, obtained by the following formula: d' = zHits = zFalseAlarms, during performance of visual search, AX-CPT and N-Back
C | 30 minutes post-intervention during both test sessions
  A measure of response bias, obtained by the following formula: C = -0.5(zHits + zFA), during performance of visual search, AX-CPT and N-Back
Checklist of Drug Related Symptoms | 1 hour post-intervention during both sessions
  Assesses physical symptoms potentially arising due to drug administration, including nausea and headache

CONTACTS AND LOCATIONS:
Overall Officials: Derek Fisher, Ph.D., Principal Investigator — Nova Scotia Health Authority
Locations (1):
- BIOTIC Neuroimaging Laboratory, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fredholm BB, Lindstrom K. Autoradiographic comparison of the potency of several structurally unrelated adenosine receptor antagonists at adenosine A1 and A(2A) receptors. Eur J Pharmacol. 1999 Sep 10;380(2-3):197-202. doi: 10.1016/s0014-2999(99)00533-6. PMID 10513579
- [Background] Ribeiro JA, Sebastiao AM. Caffeine and adenosine. J Alzheimers Dis. 2010;20 Suppl 1:S3-15. doi: 10.3233/JAD-2010-1379. PMID 20164566
- [Background] Lorist MM, Tops M. Caffeine, fatigue, and cognition. Brain Cogn. 2003 Oct;53(1):82-94. doi: 10.1016/s0278-2626(03)00206-9. PMID 14572506
- [Background] Kruger A. Chronic psychiatric patients' use of caffeine: pharmacological effects and mechanisms. Psychol Rep. 1996 Jun;78(3 Pt 1):915-23. doi: 10.2466/pr0.1996.78.3.915. PMID 8711047
- [Background] Strassnig M, Brar JS, Ganguli R. Increased caffeine and nicotine consumption in community-dwelling patients with schizophrenia. Schizophr Res. 2006 Sep;86(1-3):269-75. doi: 10.1016/j.schres.2006.05.013. Epub 2006 Jul 20. PMID 16859897
- [Background] Rogers PJ, Heatherley SV, Hayward RC, Seers HE, Hill J, Kane M. Effects of caffeine and caffeine withdrawal on mood and cognitive performance degraded by sleep restriction. Psychopharmacology (Berl). 2005 Jun;179(4):742-52. doi: 10.1007/s00213-004-2097-y. Epub 2005 Jan 26. PMID 15887055
- [Background] Ferre S, Fuxe K, von Euler G, Johansson B, Fredholm BB. Adenosine-dopamine interactions in the brain. Neuroscience. 1992 Dec;51(3):501-12. doi: 10.1016/0306-4522(92)90291-9. No abstract available. PMID 1488111
- [Background] Lucas PB, Pickar D, Kelsoe J, Rapaport M, Pato C, Hommer D. Effects of the acute administration of caffeine in patients with schizophrenia. Biol Psychiatry. 1990 Jul 1;28(1):35-40. doi: 10.1016/0006-3223(90)90429-6. PMID 2375945
- [Background] Mayo KM, Falkowski W, Jones CA. Caffeine: use and effects in long-stay psychiatric patients. Br J Psychiatry. 1993 Apr;162:543-5. doi: 10.1192/bjp.162.4.543. PMID 8481748
- [Background] Zaslove MO, Russell RL, Ross E. Effect of caffeine intake on psychotic in-patients. Br J Psychiatry. 1991 Oct;159:565-7. doi: 10.1192/bjp.159.4.565. PMID 1751869
- [Background] Carrillo JA, Benitez J. Clinically significant pharmacokinetic interactions between dietary caffeine and medications. Clin Pharmacokinet. 2000 Aug;39(2):127-53. doi: 10.2165/00003088-200039020-00004. PMID 10976659
- [Background] Odom-White A, de Leon J. Clozapine levels and caffeine. J Clin Psychiatry. 1996 Apr;57(4):175-6. No abstract available. PMID 8601555
- [Background] Koppelstaetter F, Poeppel TD, Siedentopf CM, Ischebeck A, Kolbitsch C, Mottaghy FM, Felber SR, Jaschke WR, Krause BJ. Caffeine and cognition in functional magnetic resonance imaging. J Alzheimers Dis. 2010;20 Suppl 1:S71-84. doi: 10.3233/JAD-2010-1417. PMID 20182040
- [Background] Koppelstaetter F, Poeppel TD, Siedentopf CM, Ischebeck A, Verius M, Haala I, Mottaghy FM, Rhomberg P, Golaszewski S, Gotwald T, Lorenz IH, Kolbitsch C, Felber S, Krause BJ. Does caffeine modulate verbal working memory processes? An fMRI study. Neuroimage. 2008 Jan 1;39(1):492-9. doi: 10.1016/j.neuroimage.2007.08.037. Epub 2007 Aug 31. PMID 17936643
- [Background] Foxe JJ, Morie KP, Laud PJ, Rowson MJ, de Bruin EA, Kelly SP. Assessing the effects of caffeine and theanine on the maintenance of vigilance during a sustained attention task. Neuropharmacology. 2012 Jun;62(7):2320-7. doi: 10.1016/j.neuropharm.2012.01.020. Epub 2012 Feb 2. PMID 22326943
- [Background] Brunye TT, Mahoney CR, Lieberman HR, Giles GE, Taylor HA. Acute caffeine consumption enhances the executive control of visual attention in habitual consumers. Brain Cogn. 2010 Dec;74(3):186-92. doi: 10.1016/j.bandc.2010.07.006. Epub 2010 Sep 15. PMID 20832925
- [Background] Anderson KJ, Revelle W. Impulsivity, caffeine, and proofreading: a test of the Easterbrook hypothesis. J Exp Psychol Hum Percept Perform. 1982 Aug;8(4):614-24. doi: 10.1037//0096-1523.8.4.614. PMID 6214611
- [Background] Patat A, Rosenzweig P, Enslen M, Trocherie S, Miget N, Bozon MC, Allain H, Gandon JM. Effects of a new slow release formulation of caffeine on EEG, psychomotor and cognitive functions in sleep-deprived subjects. Hum Psychopharmacol. 2000 Apr;15(3):153-170. doi: 10.1002/(SICI)1099-1077(200004)15:33.0.CO;2-C. PMID 12404329
- [Background] Lorist MM, Snel J, Kok A, Mulder G. Acute effects of caffeine on selective attention and visual search processes. Psychophysiology. 1996 Jul;33(4):354-61. doi: 10.1111/j.1469-8986.1996.tb01059.x. PMID 8753934
- [Background] Gur RE, Petty RG, Turetsky BI, Gur RC. Schizophrenia throughout life: sex differences in severity and profile of symptoms. Schizophr Res. 1996 Jul;21(1):1-12. doi: 10.1016/0920-9964(96)00023-0. PMID 8864248
- [Background] Asarnow RF, MacCrimmon DJ. Residual performance deficit in clinically remitted schizophrenics: a marker of schizophrenia? J Abnorm Psychol. 1978 Dec;87(6):597-608. doi: 10.1037//0021-843x.87.6.597. No abstract available. PMID 739083
- [Background] Kurtz MM, Ragland JD, Bilker W, Gur RC, Gur RE. Comparison of the continuous performance test with and without working memory demands in healthy controls and patients with schizophrenia. Schizophr Res. 2001 Mar 30;48(2-3):307-16. doi: 10.1016/s0920-9964(00)00060-8. PMID 11295383
- [Background] Braff DL, Light GA. The use of neurophysiological endophenotypes to understand the genetic basis of schizophrenia. Dialogues Clin Neurosci. 2005;7(2):125-35. doi: 10.31887/DCNS.2005.7.2/dlbraff. PMID 16262208
- [Background] Kahn PV, Walker TM, Williams TS, Cornblatt BA, Mohs RC, Keefe RS. Standardizing the use of the Continuous Performance Test in schizophrenia research: a validation study. Schizophr Res. 2012 Dec;142(1-3):153-8. doi: 10.1016/j.schres.2012.09.009. Epub 2012 Oct 3. PMID 23040735
- [Background] Carr VJ, Dewis SA, Lewin TJ. Preattentive visual search and perceptual grouping in schizophrenia. Psychiatry Res. 1998 Jun 15;79(2):151-62. doi: 10.1016/s0165-1781(98)00035-3. PMID 9705053
- [Background] Gold JM, Fuller RL, Robinson BM, Braun EL, Luck SJ. Impaired top-down control of visual search in schizophrenia. Schizophr Res. 2007 Aug;94(1-3):148-55. doi: 10.1016/j.schres.2007.04.023. Epub 2007 Jun 4. PMID 17544632
- [Background] Luck SJ, Gold JM. The construct of attention in schizophrenia. Biol Psychiatry. 2008 Jul 1;64(1):34-9. doi: 10.1016/j.biopsych.2008.02.014. Epub 2008 Mar 28. PMID 18374901
- [Background] Baddeley A. Working Memory: The Interface between Memory and Cognition. J Cogn Neurosci. 1992 Summer;4(3):281-8. doi: 10.1162/jocn.1992.4.3.281. PMID 23964884
- [Background] Cohen JD, Perlstein WM, Braver TS, Nystrom LE, Noll DC, Jonides J, Smith EE. Temporal dynamics of brain activation during a working memory task. Nature. 1997 Apr 10;386(6625):604-8. doi: 10.1038/386604a0. PMID 9121583
- [Background] Krieger S, Lis S, Janik H, Cetin T, Gallhofer B, Meyer-Lindenberg A. Executive function and cognitive subprocesses in first-episode, drug-naive schizophrenia: an analysis of N-back performance. Am J Psychiatry. 2005 Jun;162(6):1206-8. doi: 10.1176/appi.ajp.162.6.1206. PMID 15930072
- [Background] Lewis DA, Hashimoto T, Volk DW. Cortical inhibitory neurons and schizophrenia. Nat Rev Neurosci. 2005 Apr;6(4):312-24. doi: 10.1038/nrn1648. PMID 15803162
- [Background] Gold JM. Cognitive deficits as treatment targets in schizophrenia. Schizophr Res. 2004 Dec 15;72(1):21-8. doi: 10.1016/j.schres.2004.09.008. PMID 15531404
- [Background] de Oliveira RV, Dall'Igna OP, Tort AB, Schuh JF, Neto PF, Santos Gomes MW, Souza DO, Lara DR. Effect of subchronic caffeine treatment on MK-801-induced changes in locomotion, cognition and ataxia in mice. Behav Pharmacol. 2005 Mar;16(2):79-84. doi: 10.1097/00008877-200503000-00002. PMID 15767842
- [Background] Dall'Igna OP, Porciuncula LO, Souza DO, Cunha RA, Lara DR. Neuroprotection by caffeine and adenosine A2A receptor blockade of beta-amyloid neurotoxicity. Br J Pharmacol. 2003 Apr;138(7):1207-9. doi: 10.1038/sj.bjp.0705185. PMID 12711619
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Murd C, Aru J, Hiio M, Luiga I, Bachmann T. Caffeine enhances frontal relative negativity of slow brain potentials in a task-free experimental setup. Brain Res Bull. 2010 Apr 29;82(1-2):39-45. doi: 10.1016/j.brainresbull.2010.01.013. Epub 2010 Feb 1. PMID 20123003
- [Background] Ruijter J, De Ruiter MB, Snel J. The effects of caffeine on visual selective attention to color: an ERP study. Psychophysiology. 2000 Jul;37(4):427-39. PMID 10934901
- [Background] Lorist MM, Snel J. Caffeine effects on perceptual and motor processes. Electroencephalogr Clin Neurophysiol. 1997 May;102(5):401-13. doi: 10.1016/s0921-884x(97)95729-5. PMID 9191584
- [Background] Loke WH. Effects of caffeine on mood and memory. Physiol Behav. 1988;44(3):367-72. doi: 10.1016/0031-9384(88)90039-x. PMID 3222359
- [Background] Zahn TP, Rapoport JL. Autonomic nervous system effects of acute doses of caffeine in caffeine users and abstainers. Int J Psychophysiol. 1987 May;5(1):33-41. doi: 10.1016/0167-8760(87)90070-5. PMID 3597168
- [Background] Ghisolfi ES, Schuch A, Strimitzer IM Jr, Luersen G, Martins FF, Ramos FL, Becker J, Lara DR. Caffeine modulates P50 auditory sensory gating in healthy subjects. Eur Neuropsychopharmacol. 2006 Apr;16(3):204-10. doi: 10.1016/j.euroneuro.2005.09.001. Epub 2005 Nov 8. PMID 16278075
- [Background] Chen Y, Parrish TB. Caffeine dose effect on activation-induced BOLD and CBF responses. Neuroimage. 2009 Jul 1;46(3):577-83. doi: 10.1016/j.neuroimage.2009.03.012. Epub 2009 Mar 13. PMID 19289172
- [Background] Lorenzo-Lopez L, Amenedo E, Cadaveira F. Feature processing during visual search in normal aging: electrophysiological evidence. Neurobiol Aging. 2008 Jul;29(7):1101-10. doi: 10.1016/j.neurobiolaging.2007.02.007. Epub 2007 Mar 7. PMID 17346855
- [Background] Shah D, Impey D, Chique-Alfonzo M, Fisher D, Lorenzo-Lopez L, Knott V. Neural effects of acute nicotinic treatment on visual spatial attention in non-smokers. Pharmacol Biochem Behav. 2011 Dec;100(2):228-36. doi: 10.1016/j.pbb.2011.08.018. Epub 2011 Aug 26. PMID 21889951
- [Background] Tieges Z, Snel J, Kok A, Richard Ridderinkhof K. Caffeine does not modulate inhibitory control. Brain Cogn. 2009 Mar;69(2):316-27. doi: 10.1016/j.bandc.2008.08.001. Epub 2008 Sep 7. PMID 18782649
- [Background] Ruijter J, Lorist MM, Snel J, De Ruiter MB. The influence of caffeine on sustained attention: an ERP study. Pharmacol Biochem Behav. 2000 May;66(1):29-37. doi: 10.1016/s0091-3057(00)00229-x. PMID 10837841
- [Background] Fisher DJ, Daniels R, Jaworska N, Knobelsdorf A, Knott VJ. Effects of acute nicotine administration on behavioral and neural (EEG) correlates of working memory in non-smokers. Brain Res. 2012 Jan 6;1429:72-81. doi: 10.1016/j.brainres.2011.10.029. Epub 2011 Oct 20. PMID 22079316
- [Background] Addicott MA, Laurienti PJ. A comparison of the effects of caffeine following abstinence and normal caffeine use. Psychopharmacology (Berl). 2009 Dec;207(3):423-31. doi: 10.1007/s00213-009-1668-3. Epub 2009 Sep 24. PMID 19777214
- [Background] Giles GE, Mahoney CR, Brunye TT, Gardony AL, Taylor HA, Kanarek RB. Differential cognitive effects of energy drink ingredients: caffeine, taurine, and glucose. Pharmacol Biochem Behav. 2012 Oct;102(4):569-77. doi: 10.1016/j.pbb.2012.07.004. Epub 2012 Jul 20. PMID 22819803
- [Background] Haddock G, McCarron J, Tarrier N, Faragher EB. Scales to measure dimensions of hallucinations and delusions: the psychotic symptom rating scales (PSYRATS). Psychol Med. 1999 Jul;29(4):879-89. doi: 10.1017/s0033291799008661. PMID 10473315
- [Background] Shohet KL, Landrum RE. Caffeine consumption questionnaire: a standardized measure for caffeine consumption in undergraduate students. Psychol Rep. 2001 Dec;89(3):521-6. doi: 10.2466/pr0.2001.89.3.521. PMID 11824711
- [Background] Fisher DJ, Grant B, Smith DM, Borracci G, Labelle A, Knott VJ. Nicotine and the hallucinating brain: effects on mismatch negativity (MMN) in schizophrenia. Psychiatry Res. 2012 Apr 30;196(2-3):181-7. doi: 10.1016/j.psychres.2012.01.026. Epub 2012 Mar 16. PMID 22425471
- [Background] Fisher DJ, Knobelsdorf A, Jaworska N, Daniels R, Knott VJ. Effects of nicotine on electroencephalographic (EEG) and behavioural measures of visual working memory in non-smokers during a dual-task paradigm. Pharmacol Biochem Behav. 2013 Jan;103(3):494-500. doi: 10.1016/j.pbb.2012.09.014. Epub 2012 Sep 28. PMID 23026057